CLINICAL TRIAL: NCT06882434
Title: Holistic Integration for Healthy Longevity and Aging in Place - Establishing Full-spectrum Community-based Care System for Older People to Maintain Wellbeing Pursuing Abilities
Brief Title: Holistic Integration for Healthy Longevity and Aging in Place
Acronym: HIHOPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other); National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Superintendent, National Taiwan Univerisity Hospital Yunlin Branch, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202404065RINA
Record Dates: First submitted 2025-03-05; First posted 2025-03-18 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Decline; Sarcopenia; Depression Disorders; Nutrition Disorder; Swallowing Difficulties; Hearing Disorder; Visual Disorder; Osteoporosis; Urologic Disorders; Polypharmacy
Keywords: HIHOPE; I-COPE; dementia; depression; dysphagia; nutrition; sarcopenia; frailty; hearing disorder; visual disorder; osteoporosis; urologic disorder; polypharmacy
MeSH Terms: conditions — Cognitive Dysfunction; Sarcopenia; Nutrition Disorders; Deglutition Disorders; Hearing Disorders; Vision Disorders; Osteoporosis; Urologic Diseases; Dementia; Depression; Frailty

STUDY DESIGN:
Intervention Model Description: This study adopts a clustered randomized controlled trial (cRCT) design, where 30 community sites are randomly assigned into two groups: intervention group and control group, with a 1:2 community allocation ratio.
  To ensure balanced distribution, the randomization process involves two stratification steps:
  Community Size Stratification: Communities are first grouped based on size (≥20 participants vs. <20 participants).
  Urban-Rural Stratification: Communities are further stratified based on their urban or rural development status.
  Within each stratum, communities are randomly allocated to the intervention or control group.
Masking Description: This study is non-blinded, meaning both participants and researchers are aware of the assigned intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The HI-HOPE Project implements a three-phase intervention over 48 weeks, integrating cognitive, physical, and social engagement strategies.
  Phase 1 (12 Weeks): Focuses on cognitive stimulation, depression relief, and music-based movement therapy. Includes weekly high-intensity exercise (3 hours/week).
  Phase 2 (12 Weeks): Covers all six ICOPE domains with community-led wellness sessions and weekly high-intensity exercise (3 hours/week).
  Phase 3 (12 Weeks): Intensive strength and mobility training (2 hours/week).
  Referral Process: Individuals with abnormal screenings receive personalized support, including transportation aid, financial assistance, telehealth, and group referrals.
  Digital Health: Uses telehealth consultations, medication tracking, and nutritional assessments to enhance care access and monitor intervention outcomes.
  Interventions: Behavioral: Local intervention program; Behavioral: Referral Process; Behavioral: Telehealth Education & Digital Integration
- Control (No Intervention): Participants in the control group will undergo the same baseline and follow-up assessments as the intervention group. After evaluation, they will be informed of any abnormal findings and provided with recommendations for appropriate medical referrals based on standard care practices.
  However, no additional referral assistance, intervention programs, or follow-up services will be provided beyond the basic healthcare guidance currently available in the community.

INTERVENTIONS:
Behavioral: Local intervention program — HI-HOPE Project introduces a three-phase intervention program Phase 1: "Active Mind & Body" (12 Weeks) Focus: Cognitive enhancement, depression relief, and music-based movement therapy.
  Delivery: Certified community instructors. Schedule: 1 session/week, 2 hours per session (total 12 sessions). Supplementary Exercise: High-intensity training by professional coaches (1 session/week, 1 hour per session).
  Phase 2: "Complete Senior Wellness" (12 Weeks) Focus: Comprehensive functional improvement covering all six ICOPE domains. Delivery: Certified community instructors. Schedule: 1 session/week, 2 hours per session (total 12 sessions). Supplementary Exercise: High-intensity training by professional coaches (1 session/week, 1 hour per session).
  Phase 3: "Advanced Exercise Training" (12 Weeks) Focus: Strengthening self-care abilities and increasing acceptance of medical interventions.
  Delivery: Professional exercise coaches. Schedule: 2 sessions/week, 1 hour per session (total 24 sessions).
  Arms: Intervention
Behavioral: Referral Process — Self-referral tracking (1-2 weeks): Participants able to visit referral sites independently will be followed up to confirm completion.
  Barrier assessment: If unable to attend, interviews will identify obstacles (e.g., transport, finances, willingness).
  Transportation support: Solutions include volunteer transport with fuel subsidies, local transport networks, and government-assisted group referrals.
  Financial assistance: Eligibility for social welfare aid will be assessed, with support for applications.
  Personal willingness & health literacy: Health education will address concerns about treatment or social stigma.
  Telehealth consultations: Remote specialist consultations will be provided if in-person visits are not possible.
  Hospital-based referral support: Group hospital visits will be arranged for those with referral difficulties.
  Monthly tracking: Referral completion rates and outcomes will be monitored (e.g., treatments, assistive devices, social services).
  Arms: Intervention
Behavioral: Telehealth Education & Digital Integration — Live-streamed health education across multiple community sites.
  Digital health platforms for real-time intervention monitoring and professional feedback:
  Polypharmacy management via medication usage tracking and pharmacist analysis. Nutritional assessment with dietitian recommendations. Health consultations provided remotely by specialists based on screening results.
  Arms: Intervention

SUMMARY:
Background:

Taiwan is experiencing rapid population aging, with a growing prevalence of chronic diseases and functional impairments among older adults. Existing Integrated Care for Older People (ICOPE) programs focus primarily on screening but lack sufficient follow-up and intervention. In response, the HI-HOPE Project was developed to establish a community-based, multidisciplinary intervention model to enhance intrinsic capacity and promote healthy aging in rural elderly populations.

Survey and Screening:

The study will be conducted in 30 community centers across Yunlin County, targeting older adults aged ≥55 years. Participants will undergo biannual screenings over two years, assessing cognitive function, depression, mobility, vitality (nutrition), hearing, vision, osteoporosis, polypharmacy, urological health, and social participation & welfare.

Intervention:

Participants will be randomly assigned to either:

HI-HOPE Integrated Care Group:

On-Site Community Interventions: Exercise training, mindfulness, social activities, oral and swallowing rehabilitation, hearing and vision training.

Telehealth & Remote Education: Digital health monitoring, remote consultations, and health education.

Referral Services: Access to specialized medical care, transportation assistance, and follow-up support.

Control Group: Standard community care services without additional structured interventions.

Outcome Measures:

Primary outcomes include changes in intrinsic capacity of functional health metrics, including abnormalities of I-COPE components (mobility, cognitive status, depression, hearing, vision, vitality) . Secondary outcomes assess quality of life, activities of daily living, hospitalization, emergency visits, falls, and mortality rates over two years.

Significance:

This project integrates digital health technologies, interdisciplinary care, and community-based interventions to improve elderly health outcomes. The findings will guide the future scalability of integrated aging care models in Taiwan and beyond.

DETAILED DESCRIPTION:
General Introduction As the population ages, the prevalence of chronic diseases and functional impairments is increasing. Since 1980, the proportion of people aged 65 and older in Taiwan has been steadily rising, and in 2018, Taiwan officially became an aged society. It is projected to reach the status of a super-aged society by 2025. Achieving healthy longevity is a shared goal in an aging society. According to the World Health Organization (WHO), the purpose of promoting healthy aging is to help older adults maintain their physical functions, allowing them to engage in activities that bring them happiness. Maintaining intrinsic capacity is a key aspect of this goal. However, many elderly individuals experience multiple chronic diseases and polypharmacy, physical decline, reduced cognitive and learning abilities, and socio-economic disadvantages. These factors contribute to the progressive deterioration of their intrinsic capacity, posing significant challenges to achieving healthy aging.

Since 2018, National Taiwan University Hospital Yunlin Branch has actively reached out to remote rural communities, providing high-quality and convenient medical and health services to the elderly in Yunlin County. Observations over the years have shown that the prevalence of metabolic syndrome among the elderly in rural Yunlin is significantly high. Nutritional imbalances have led to 35.35% of elderly individuals having a BMI above the normal range, while 48.4% have stage II hypertension. Sarcopenia is also a concerning issue: 50.36% of seniors exhibit low grip strength, 16.82% require more than 16 seconds to complete five sit-to-stand movements, and 77.92% show signs of lower limb weakness in a 3-meter walk test. Compared to other regions in Taiwan and internationally, the elderly in Yunlin demonstrate lower physical fitness levels, highlighting the need for greater attention and assistance in ensuring their health and well-being.

Currently, a person-centered, community-based, integrated multidisciplinary assessment and intervention approach is the mainstream method for promoting health among older adults, supported by international evidence. The Integrated Care for Older People (ICOPE) model, proposed by the World Health Organization (WHO), identifies six key intrinsic capacities that need to be maintained for healthy aging: cognition, mobility, nutrition, depression, hearing, and vision. In 2017, WHO published community-level intervention guidelines that provided detailed assessments and recommendations for integrated community-based care. The guidelines emphasize resource integration, follow-up interventions, and a well-structured healthcare support system to enhance community-wide care.

The Health Promotion Administration (HPA) of Taiwan's Ministry of Health and Welfare has actively promoted the ICOPE framework. In 2021, it launched a pilot program for assessing and preventing functional decline in older adults, led by local health departments. By 2023, this initiative had expanded to all 22 counties and cities across Taiwan, with hospitals and medical institutions collaborating to conduct screenings. However, the current ICOPE implementation model is still primarily hospital-centered, making it less accessible to older adults in remote or mobility-limited communities.

A literature review and expert discussions indicate that Taiwan's ICOPE model focuses mainly on screening, with insufficient follow-up and referral systems. Due to the diverse and complex health issues faced by older adults, implementing follow-up care remains a major challenge. For example, in Yunlin County, nearly 8,000 screening surveys were completed in 2022, yet half of those who needed follow-up assessments did not receive referrals, and 95% of cases lacked follow-up within six months. Despite significant efforts by Yunlin's health authorities to implement ICOPE, the lack of case management personnel and a comprehensive medical support system has made intervention and follow-up care difficult. Thus, establishing a structured intervention model and improving implementation strategies is crucial for the future development of ICOPE in Taiwan.

Currently, various health promotion programs operate independently, often lacking sufficient cross-sector communication. This results in low service utilization rates due to unclear resource availability for elderly individuals and caregivers. Different approaches to community-based elderly care-such as hospital referrals, on-site community interventions, and telehealth monitoring-should be integrated to provide the most appropriate care and support.

To address these challenges, National Taiwan University Hospital Yunlin Branch is leveraging its experience in the Apollo Community Care Model, in collaboration with The National Health Research Institutes Aging and Health Welfare Research Center, The Yunlin County Government, and Yunlin University of Science and Technology. This initiative introduces the HI-HOPE Project, which focuses on

A senior-centered, community-based model A ten-core functional assessment and intervention strategy Integrated medical and digital health resources Interdisciplinary collaboration to enhance elderly well-being

The HI-HOPE Project builds upon existing community-based elderly care programs, particularly the pharmaceutical care model for polypharmacy management and the osteoporosis and sarcopenia risk assessment project in Yunlin County. Using these programs as a foundation, HI-HOPE will implement clustered randomized controlled trials (RCTs) across 30 community sites in Yunlin County, targeting older adults aged 55 and above. The project will establish two groups, including HI-HOPE Integrated Care Group (10 communities) and Control Group (20 communities). The HI-HOPE group expands upon WHO's ICOPE six dimensions, adding osteoporosis, polypharmacy, urological health, and social welfare, creating a comprehensive ten-core framework. Social welfare services will integrate existing government programs such as cancer screening, digital health, and long-term care resources.

The intervention model consists of three primary components:

On-Site Community Interventions - Including exercise training, mindfulness meditation, social participation activities, oral and swallowing rehabilitation, hearing rehabilitation, and vision training.

Telehealth and Remote Education - Leveraging digital technologies for health education, monitoring, and consultations.

Referral Services - Facilitating access to medical care, transportation assistance, and follow-up support.

The project will run for two years, with biannual screenings to track changes in intrinsic capacity, core health functions, and life events, such as falls, fractures, emergency visits, hospitalizations, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥55 years (includes older adults and pre-elderly individuals).
* No severe functional disability (must be able to walk independently, use assistive devices, or operate a wheelchair independently).
* No severe cognitive impairment (must be able to respond appropriately to verbal questions).

Exclusion Criteria:

* Irregular community participation (less than once per week in the target community).
* Mild dementia or greater (assessed during screening). If identified, family members will be notified, and they retain the right to withdraw the participant unconditionally.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Intrinsic capacity | The primary outcome (intrinsic capacity) will be assessed every six months over a two-year period, totaling four evaluations throughout the study duration.
  The primary outcome is intrinsic capacity, measured by the total number of impaired ICOPE (Integrated Care for Older People) domains (0-6). Impairment criteria are: (1) Cognitive: Mini-Mental State Examination (MMSE) <24; (2) Depression: Geriatric Depression Scale (GDS-15) >6; (3) Mobility: Short Physical Performance Battery (SPPB) ≤9; (4) Vitality: Mini Nutritional Assessment-Short Form (MNA-SF) ≤11; (5) Vision: ICOPE-WHO Simple Vision Test abnormal if failing distance/near vision tests or having an eye disease/chronic condition (e.g., diabetes, hypertension) without an eye exam in the past year; (6) Hearing: ICOPE Whispered Voice Test abnormal. Each domain is assessed separately and classified as either impaired (0) or not impaired (1) based on the predefined criteria. The final intrinsic capacity score is the sum of non-impaired domains (range: 0-6), with higher scores indicating greater intrinsic capacity.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Every 6 months, for 2 years
  Score change in Mini-Mental State Examination (MMSE), range 0-30, lower score indicates higher abnormality.
Brain Health Test (BHT) | Every 6 months, for 2 years
  Score change in Brain Health Test (BHT), range 0-28, lower score indicates higher abnormality.
Geriatric Depression Scale-15 (GDS-15) | Every 6 months, for 2 years
  Score change in Geriatric Depression Scale-15 (GDS-15), range 0-15, higher score indicates more severe depressive symptoms.
Geriatric Anxiety Inventory (GAI) | Every 12 months, for 2 years
  Score change in Geriatric Anxiety Inventory (GAI), range 0-20, higher score indicates more severe anxiety symptoms.
Chinese Happiness Inventory (CHI) | Every 12 months, for 2 years
  Score change in Chinese Happiness Inventory (CHI), range 0-100, higher score indicates greater subjective well-being.
Handgrip Strength | Every 6 months, for 2 years
  Change in Handgrip Strength Test, measured in kilograms (kg), lower score indicates reduced muscle strength.
Short Physical Performance Battery (SPPB) | Every 6 months, for 2 years
  Score change in Short Physical Performance Battery (SPPB), range 0-12, lower score indicates poorer physical performance.
Appendicular Skeletal Muscle Index (ASMI) | Every 6 months, for 2 years
  Score change in Appendicular Skeletal Muscle Index (ASMI), measured in kg/m², lower score indicates lower muscle mass.
International Physical Activity Questionnaire (IPAQ) | Every 6 months, for 2 years
  Score change in International Physical Activity Questionnaire (IPAQ), measured in MET-minutes/week, lower score indicates lower physical activity level.
Mini Nutritional Assessment-Short Form (MNA-SF) | Every 6 months, for 2 years
  Score change in Mini Nutritional Assessment-Short Form (MNA-SF), range 0-14, lower score indicates higher risk of malnutrition.
Body Mass Index (BMI) | Every 6 months, for 2 years
  Score change in Body Mass Index (BMI), measured in kg/m², lower or higher values outside normal range (18.5-24.9 kg/m²) indicate underweight or overweight/obesity, respectively.
Oral Frailty Assessment Scale (OF-5) | Every 12 months, for 2 years
  Score change in Oral Frailty Assessment Scale (OF-5), range 0-5, higher score indicates greater oral frailty and functional decline.
Community Periodontal Index (CPI) score | Every 12 months, for 2 years
  Score change in Community Periodontal Index (CPI) score, range 0-4, higher score indicates worse periodontal status.
Loss of Attachment (LA) code | Every 12 months, for 2 years
  Score change in Loss of Attachment (LA) code, range 0-4, higher score indicates more severe periodontal attachment loss.
Decayed, Missing, and Filled Teeth (DMFT) | Every 12 months, for 2 years
  Change in number of Decayed, Missing, and Filled Teeth (DMFT), total count of affected teeth, higher number indicates worse dental caries history and oral health status
Tongue base ultrasonography | Every 12 months, for 2 years
  Ultrasonographic measurement of mylohyoid muscle thickness(mm), cross-sectional area of geniohyoid muscle (mm²), cross-sectional area of genioglossus muscle (mm²), total thickness from chin base to tongue upper surface, (mm). Lower value may indicate reduced structural support related to swallowing and speech functions.
Hearing Handicap Inventory for the Elderly - Short Form, Chinese version (HHIE-C) | Every 12 months, for 2 years
  Score change in Hearing Handicap Inventory for the Elderly - Short Form, Chinese version (HHIE-C), range 0-40, higher score indicates greater perceived hearing handicap.
International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI-SF) | Every 12 months, for 2 years
  Score change in International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI-SF), range 0-21, higher score indicates greater severity of urinary incontinence and impact on quality of life.
EuroQol-5 Dimension 5-Level (EQ-5D-5L) | Every 6 months, for 2 years
  Score change in EuroQol-5 Dimension 5-Level (EQ-5D-5L) index score, standarized range -1 to 1, higher score indicates better health-related quality of life.
Barthel Index (for activities of daily living) | Every 6 months, for 2 years
  Score change in Barthel Index (for activities of daily living), range 0-100, higher score indicates greater independence in basic activities of daily living
Instrumental Activities of Daily Living (IADL) | Every 6 months, for 2 years
  Score change in Instrumental Activities of Daily Living (IADL), range 0-8, higher score indicates greater independence in performing instrumental daily tasks.
Health Events | Every 3 months, for 2 years
  Numbers of falls, fractures, emergency visits, hospitalizations, institutionalization, and mortality tracking.
Fracture Risk Assessment Tool (FRAX) | Before the intervention (baseline) and at 24th month
  Score change in Fracture Risk Assessment Tool (FRAX), estimated 10-year probability (%) of major osteoporotic fractures and hip fractures, higher percentage indicates greater fracture risk.
Bone Mineral Density (BMD) | Before the intervention (baseline) and at 24th month
  Score change in Dual-energy X-ray Absorptiometry (DXA), measured as Bone Mineral Density (BMD) in g/cm² and T-score, lower BMD or T-score indicates higher risk of osteoporosis.
Polypharmacy | Every 6 months, for 2 years
  Number of currently used drugs, total count, higher number indicates polypharmacy risk.
Anticholinergic burden (ACB) | Every 6 months, for 2 years
  Anticholinergic burden, cumulative score (0-3) based on medications with anticholinergic properties from reviewed literatures, higher score indicates greater risk of cognitive and physical side effects.
Potentially Inappropriate Medications (PIMs) | Every 6 months, for 2 years
  Number of Potentially Inappropriate Medications (PIMs), total count based on established criteria, higher number indicates greater prescribing risk.
Number of drugs with fall risk | Every 6 months, for 2 years
  Total count of medications associated with increased fall risk
Number of drug-related problems (DRPs) | Every 6 months, for 2 years
  Total identified issues according to The Pharmaceutical Care Network Europe (PCNE), including drug interactions, duplications, inappropriate dosing, higher count indicates greater pharmacotherapy risk.
ARMS (Adherence to Refills and Medications Scale) | Every 6 months, for 2 years
  ARMS (Adherence to Refills and Medications Scale) is a validated questionnaire designed to assess how well individuals adhere to their prescribed medication and refill schedules. It consists of 12 questions (range 12-48), with lower scores indicating better adherence to medication and higher scores suggesting potential issues with adherence.

OTHER OUTCOMES:
Ishihara Color Blindness Test | Every 12 months, for 2 years
  Abnormality by Ishihara Color Blindness Test (yea/no)
AMSLER Grid | Every 12 months, for 2 years
  AMSLER Grid, measured as presence (yes/no) of visual distortion or scotoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Ang S. Social participation and health over the adult life course: Does the association strengthen with age? Soc Sci Med. 2018 Jun;206:51-59. doi: 10.1016/j.socscimed.2018.03.042. Epub 2018 Apr 14. PMID 29684648
- [Background] Blancafort Alias S, Cuevas-Lara C, Martinez-Velilla N, Zambom-Ferraresi F, Soto ME, Tavassoli N, Mathieu C, Heras Muxella E, Garibaldi P, Anglada M, Amblas J, Santaeugenia S, Contel JC, Domingo A, Salva Casanovas A. A Multi-Domain Group-Based Intervention to Promote Physical Activity, Healthy Nutrition, and Psychological Wellbeing in Older People with Losses in Intrinsic Capacity: AMICOPE Development Study. Int J Environ Res Public Health. 2021 Jun 2;18(11):5979. doi: 10.3390/ijerph18115979. PMID 34199566
- [Background] Cheng YC, Kuo YC, Chang PC, Li YC, Huang WT, Chen W, Chou CY. Geriatric Functional Impairment Using the Integrated Care for Older People (ICOPE) Approach in Community-Dwelling Elderly and Its Association with Dyslipidemia. Vasc Health Risk Manag. 2021 Jul 5;17:389-394. doi: 10.2147/VHRM.S305490. eCollection 2021. PMID 34262283
- [Background] Rojano I Luque X, Blancafort-Alias S, Prat Casanovas S, Forne S, Martin Vergara N, Fabregat Povill P, Vila Royo M, Serrano R, Sanchez-Rodriguez D, Vilchez Saldana M, Martinez I, Dominguez Lopez M, Riba Porquet F, Intxaurrondo Gonzalez A, Salva Casanovas A. Identification of decreased intrinsic capacity: Performance of diagnostic measures of the ICOPE Screening tool in community dwelling older people in the VIMCI study. BMC Geriatr. 2023 Feb 21;23(1):106. doi: 10.1186/s12877-023-03799-0. PMID 36809987
- [Background] Chew J, Lim JP, Yew S, Yeo A, Ismail NH, Ding YY, Lim WS. Disentangling the Relationship between Frailty and Intrinsic Capacity in Healthy Community-Dwelling Older Adults: A Cluster Analysis. J Nutr Health Aging. 2021;25(9):1112-1118. doi: 10.1007/s12603-021-1679-2. PMID 34725670
- [Background] Zhao J, Chhetri JK, Chang Y, Zheng Z, Ma L, Chan P. Intrinsic Capacity vs. Multimorbidity: A Function-Centered Construct Predicts Disability Better Than a Disease-Based Approach in a Community-Dwelling Older Population Cohort. Front Med (Lausanne). 2021 Sep 28;8:753295. doi: 10.3389/fmed.2021.753295. eCollection 2021. PMID 34651003
- [Background] Prince MJ, Acosta D, Guerra M, Huang Y, Jacob KS, Jimenez-Velazquez IZ, Jotheeswaran AT, Llibre Rodriguez JJ, Salas A, Sosa AL, Acosta I, Mayston R, Liu Z, Llibre-Guerra JJ, Prina AM, Valhuerdi A. Intrinsic capacity and its associations with incident dependence and mortality in 10/66 Dementia Research Group studies in Latin America, India, and China: A population-based cohort study. PLoS Med. 2021 Sep 14;18(9):e1003097. doi: 10.1371/journal.pmed.1003097. eCollection 2021 Sep. PMID 34520466
- [Background] Gonzalez-Bautista E, de Souto Barreto P, Andrieu S, Rolland Y, Vellas B; MAPT/DSA group (members are listed under 'Contributors'). Screening for intrinsic capacity impairments as markers of increased risk of frailty and disability in the context of integrated care for older people: Secondary analysis of MAPT. Maturitas. 2021 Aug;150:1-6. doi: 10.1016/j.maturitas.2021.05.011. Epub 2021 Jun 4. PMID 34274071
- [Background] Lu F, Li J, Liu X, Liu S, Sun X, Wang X. Diagnostic performance analysis of the Integrated Care for Older People (ICOPE) screening tool for identifying decline in intrinsic capacity. BMC Geriatr. 2023 Aug 23;23(1):509. doi: 10.1186/s12877-023-04180-x. PMID 37612657
- [Background] Leung AYM, Su JJ, Lee ESH, Fung JTS, Molassiotis A. Intrinsic capacity of older people in the community using WHO Integrated Care for Older People (ICOPE) framework: a cross-sectional study. BMC Geriatr. 2022 Apr 8;22(1):304. doi: 10.1186/s12877-022-02980-1. PMID 35395736
- [Background] Chang KC, Hung SH, Hsueh SJ, Chao SF, Huang WL, Chen HS, Jeng Y, Chen HH, Hwang JJ, Liou HH. Development of the Houston-Apollo model for older people living in remote areas in Taiwan. Geriatr Gerontol Int. 2021 Mar;21(3):299-305. doi: 10.1111/ggi.14130. Epub 2021 Feb 1. PMID 33527540